CLINICAL TRIAL: NCT05340166
Title: Comparative Evaluation of the Ultrasound-guided Radiofrequency Neurolysis and Chemical Neurolysis of the Genicular Nerves
Brief Title: Evaluation of Radiofrequency Neurolysis and Chemical Neurolysis of the Genicular Nerves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, Principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 131/01
Record Dates: First submitted 2022-04-14; First posted 2022-04-22 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiofrequency Neurolysis (Active Comparator): Radiofrequency Neurolysis of genicular nerves
  Interventions: Procedure: Genicular nerve radiofrequency neurolysis
- Chemical Neurolysis (Experimental): Chemical Neurolysis of genicular nerves
  Interventions: Procedure: Genicular nerve chemical neurolysis

INTERVENTIONS:
Procedure: Genicular nerve radiofrequency neurolysis — Neurolysis of superomedial, superolateral and inferomedial genicular nerves
  Arms: Radiofrequency Neurolysis
Procedure: Genicular nerve chemical neurolysis — Neurolysis of superomedial, superolateral and inferomedial genicular nerves
  Arms: Chemical Neurolysis

SUMMARY:
Knee osteoarthritis is one of the most common causes of pain and loss of function in the elderly population and is a source of socioeconomic costs. Selective denervation of the superior medial, superior lateral and inferior medial genicular nerves, which provide the sensory innervation of the knee joint, is an effective treatment method used to relieve pain and improve functional capacity. Radiofrequency neurolysis of genicular nerves (RFN) is accepted as an effective technique for the treatment of knee pain. However, due to higher equipment costs, longer procedure times, and procedure-related pain, alternative treatments are needed.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Coagulation disorders
* Rheumatoid disorders
* Infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-24 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Change from baseline to 6 months after procedure
  Pain Score Change The 11-point NRS consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The patient is instructed to identify one number between 0 and 10, which is best representative of their pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: selin guven kose, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)